CLINICAL TRIAL: NCT02804555
Title: Effects of Intraoperative Oxygen Therapy on Oxygenation and Reactive Oxygen Species Levels of Newborns Born Via Elective Cesarian Section
Brief Title: Effects of Intraoperative Oxygen Therapy on Oxygenation of Newborns Born Via Elective Cesarian Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Domonkos Trásy, clinician, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Maternal hyperoxia
Record Dates: First submitted 2016-06-06; First posted 2016-06-17 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2016-11

CONDITIONS: Obstetrical Complication of Anesthesia
Keywords: reactive oxygen species; elective cesarean section; oxygen therapy; newborn
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen support (Active Comparator): 5 liter / minute oxygen has given to the mothers on face mask.
  Interventions: Other: Oxygen
- Room air (No Intervention): Oxygen support has not given to the mothers.

INTERVENTIONS:
Other: Oxygen — Oxygen administration
  Arms: Oxygen support

SUMMARY:
In this study the investigators examine the effects of intraoperative oxygen administration to the mother on certain enzyme functions of the newborn. With this object blood samples are taken from the newborn's umbilical chord - which is otherwise a routine practice at the investigators clinic - and the mother's radial artery in parallel with umbilical clamping and cutting for blood gas and reactive oxygen species analyses. Samples are analyzed locally in a properly equipped laboratory.

DETAILED DESCRIPTION:
Whole-blood superoxide and hydrogen peroxide production was measured from the newborn's umbilical chord.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section.
* Signed informed consent form.

Exclusion Criteria:

* Subject meets the definition of a vulnerable subject as defined in International Organization for Standardization 14155:2011.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Hyperoxia Newborns | through study completion up to two years
  We measured umbilical vein blood gas parameters.

SECONDARY OUTCOMES:
Maternal hyperoxia | through study completion up to two years
  We measured arterial blood gas parameters of the mother from radial artery.
Alterations in newborns' enzyme functions due to maternal hyperoxia | through study completion up to two years
  We measured umbilical vein reactive oxygen species (ROS) of the newborn.

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Molnar, MD, Principal Investigator — Szeged University
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Undecided